CLINICAL TRIAL: NCT04085835
Title: Evolution and Genetic Basis of Menstruation in Women
Brief Title: Evolution of Menstruation
Acronym: EVOMENS
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C18-19; 2019-A01089-48 (Registry Identifier: INSERM)
Record Dates: First submitted 2019-09-05; First posted 2019-09-11 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Menstruation
Keywords: endometrium; comparative genomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Uterine lining (endometrium) samples obtained from menstrual fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study examines gene expression and gene regulation in the uterine lining during menses in women, for evolutionary comparison with other primates which do or do not menstruate. Samples will be obtained by non-invasive collection of menstrual fluid from healthy donors.

DETAILED DESCRIPTION:
Menstruation corresponds to the shedding of the uterine lining when fecundation has not occurred. This is a recent evolutionary innovation in primates, and the cellular and genetic changes that led to the acquisition of menstruation are not well understood. Additionally, the uterine lining is poorly characterized in humans at the menstrual time point, which hinders both evolutionary and medically-relevant analyses.

In this study, the research team are collecting menstrual fluid samples from healthy female volunteers to profile gene expression and gene regulatory elements in the major cell types that compose the uterine lining during menstruation. The investigators will compare this data to similar samples collected from other primates at the same time point in the female hormonal cycle.

The objective is to identify genes that have acquired novel regulation and/or expression patterns and which may be involved in menstruation.

ELIGIBILITY:
Inclusion Criteria:

* having regular periods
* being comfortable using silicone menstrual hygiene devices ("cup")
* having giving consent in writing

Exclusion Criteria:

* use of an internal contraception method (hormone or non-hormone based) during or within three months before the study
* pregnancy during or within three months before the study
* amenorrhea (absent periods) during or within three months before the study
* gynaecological intervention or surgery within three months before the study
* hormonal treatment during or within three months before the study
* absence of written consent
* breastfeeding
* medical treatment during the study
* low (< 18.5) or high (> 30) body mass index (BMI)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy female volunteers experiencing regular periods
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2025-04-27 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
Gene expression levels measured by RNA-seq | Average to study completion 30 months
  Gene expression levels measured in the different cell types of the endometrial tissue during menstruation using RNA extraction and sequencing (RNA-seq)
Active regulatory elements profiled by ATAC-seq | Average to study completion 30 months
  Profiling of the genetic elements accessible to transposase assays and sequencing (putative active regulatory elements; ATAC-seq) in the different cell types of endometrial tissue during menstruation

CONTACTS AND LOCATIONS:
Overall Officials: Camille Berthelot, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Institut de Biologie de l'Ecole Normale Superieure, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided